CLINICAL TRIAL: NCT04457063
Title: Endothelial Cell Loss Following Toric ICL Implantation for Correction of Myopia and Astigmatism After Penetrating Keratoplasty
Brief Title: Endothelial Cell Loss After Penetrating Keratoplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0304624
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: A prospective non-comparative non-randomized clinical study which was conducted on 12 eyes of 8 patients 4 males and 4 females who underwent PKP for keratoconus, and then toric ICL was implanted after minimum of one year with stable refraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- penetrating keratoplasty (Experimental): A prospective non-comparative non-randomized clinical study which was conducted on 12 eyes of 8 patients 4 males and 4 females who underwent PKP for keratoconus, and then toric ICL was implanted after minimum of one year with stable refraction
  Interventions: Procedure: PKP

INTERVENTIONS:
Procedure: PKP — 1. The horizontal axis was marked with a pointed marker at the slit lamp immediately before surgery.
  2. TICL loading into the STAAR injector cartridge
  3. Temporal clear corneal 3 mm incision & 2-side ports then viscoelastic injection into the AC
  4. Implantation of the TICL using the injector, then rotation according to the implantation diagram guided with Mendez protractor, and lastly placement of the haptics under the iris.
  5. Pupil constriction with A.Ch.
  6. Washing the viscoelastic &Wound hydration.
  7. Topical antibiotic steroids (Vigamox and Tobradex) 4 times /day for 3weeks

SUMMARY:
This work aimed at the assessment of corneal endothelial cell loss after toric ICL implantation for correction of myopia and astigmatism after penetrating keratoplasty.

DETAILED DESCRIPTION:
Penetrating keratoplasty (PKP) is considered a safe and effective procedure.This work aimed at the assessment of corneal endothelial cell loss after toric ICL implantation for correction of myopia and astigmatism after penetrating keratoplasty.

ELIGIBILITY:
Inclusion Criteria:

* PKP for keratoconus, and then toric ICL was implanted after minimum of one year with stable refraction

Exclusion Criteria:

* Less than 18 and unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Refraction | 1 year
  Refractive measured by Diopter
Visual acuity | 1 year
  The decimal snellens
Intra-ocular pressure | 1 year
  mg

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Mossallam, PhD, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No